CLINICAL TRIAL: NCT04418505
Title: A Randomized Study Evaluating the Efficacy of the Vielight RX Plus in the Treatment of COVID-19 Respiratory Symptoms
Brief Title: Vielight RX Plus for the Treatment of COVID-19 Respiratory Symptoms
Acronym: COVIDLight
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vielight Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VL-2020-02
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-CoV-2; Photobiomodulation; Low level light therapy; PBM; Red light; Near-infrared light; At-home treatment; Remote
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Prospective, randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (No Intervention): This group will not receive Vielight RX Plus treatment. Instead, they will follow the COVID-19 standard of treatment recommended by Health Canada.
- Standard of Care + Vielight RX Plus Treatment (Experimental): The is group will receive Vielight RX Plus treatment and follow the COVID-19 standard of treatment recommended by Health Canada.
  Interventions: Device: Vielight RX Plus

INTERVENTIONS:
Device: Vielight RX Plus — The Vielight RX Plus is designed to deliver near-infrared light and red light via LEDs placed directly on the manubrium of the sternum (which covers the thymus gland) and inside one nostril, respectively.
  Arms: Standard of Care + Vielight RX Plus Treatment

SUMMARY:
The objective of this study is to obtain data on the efficacy of the Vielight RX Plus in decreasing time to recovery of symptoms in subjects with COVID-19. The study will be conducted among COVID-19 positive subjects at home in self-isolation via electronic data collection (EDC). There will be no physical contact between the subjects and the Qualified Investigator (QI) or other study staff. This study aims to demonstrate that the Vielight RX Plus is a useful adjunct to standard of care (SOC). We hypothesize that the Vielight RX Plus will accelerate recovery and reduce viral infection severity.

DETAILED DESCRIPTION:
This study is conducted entirely online. At no point will study staff be in direct contact with participants. The study will be managed by an independent clinical research organization (CRO), supporting a Qualified Investigator (QI). Vielight Inc will supply the RX Plus devices free of charge and will sponsor the study.

Potential participants will be prompted to complete an online screening form if they are interested in participating. During the screening, the potential participant will be asked to upload a copy of their positive COVID-19 infection confirmation report and a valid ID. If the potential subject qualifies for the study, by statisfying all inclusion and exclusion criteria, the potential participant will then be prompted to complete an electronic informed consent form (ICF) via the electronic data collection (EDC) platform and will be enrolled into the study.

This is a 30-day, prospective, randomized study, with no blinding. 280 participants will be randomized into two groups: Group 1: Standard of Care; Group 2: Standard of Care + Vielight RX Plus treatment. In Group 2, the Vielight RX Plus will be administered for 20 minutes twice a day, separated by at least 6 hours for the first 5 days. For the subsequent 25 days, treatment will be once per day. The Vielight RX Plus will be positioned over the upper most part of the breastbone to stimulate the thymus gland and within one nostril.

During each of the 30-days, participants will be asked to complete a questionnaire to assess respiratory symptom severity, and log a daily dairy as well as oxygen saturation level (using a portable oximeter).

The primary measure is time to overall recovery in days.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of COVID-19 infection
* Experiencing moderate to severe respiratory symptoms
* Between 18-65 years of age

Exclusion Criteria:

* Need for hospitalization at the time of diagnosis
* Current need for supplemental oxygen or positive pressure support and/or has required supplemental oxygen or positive pressure support for >or= 24 hours
* >10 days since symptom onset
* Diagnosis of Chronic Obstructive Pulmonary Disease (COPD)
* Pregnant
* Positive for Hepatitis C Virus (HCV), Hepatitis B Virus (HBV) or Human Immunodeficiency Virus
* Inability to electronically complete study questionnaires in English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Time to recovery | 30 days

SECONDARY OUTCOMES:
Time to elimination of COVID-19 related symptoms | 30 days
Mean number of days with mild COVID-19 related symptoms | 30 days
Mean number of days with mild overall respiratory symptoms | 30 days
Time to symptom reduction | 30 days
Time to elimination of symptoms | 30 days
Average number of days with mild respiratory symptoms | 30 days
Oxygen saturation | 30 days
Hospitalization rate | 30 days
Mortality | 30 days

CONTACTS AND LOCATIONS:
Locations (2):
- Progressive Medical Research, Port Orange, Florida, United States
- Dr. Michael Zahavi, Oshawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lim L, Hosseinkhah N, Van Buskirk M, Berk A, Loheswaran G, Abbaspour Z, Karimpoor M, Smith A, Ho KF, Pushparaj A, Zahavi M, White A, Rubine J, Zidel B, Henderson C, Clayton RG, Tingley DR, Miller DJ, Karimpoor M, Hamblin MR. Photobiomodulation Treatment with a Home-Use Device for COVID-19: A Randomized Controlled Trial for Efficacy and Safety. Photobiomodul Photomed Laser Surg. 2024 Jun;42(6):393-403. doi: 10.1089/pho.2023.0179. Epub 2024 Jun 19. PMID 38940733